CLINICAL TRIAL: NCT07080905
Title: Phase 3, Open-label, Single-dose, Multicenter Study Investigating Efficacy, Safety, and Tolerability of CSL222 (Etranacogene Dezaparvovec) Administered to Adolescent Male Subjects (≥ 12 to < 18 Years of Age) With Severe or Moderately Severe Hemophilia B
Brief Title: Phase 3, Open-label, Single-dose Study of CSL222 in Adolescent Male Subjects (≥ 12 to < 18 Years of Age) With Severe or Moderately Severe Hemophilia B
Acronym: IX-TEND 3004
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSL222_3004; 2023-505805-18-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-07; First posted 2025-07-23 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- CSL222 (Experimental): Participants will receive CSL222 as a single intravenous (IV) infusion of 2 × 10^13 genome copies per kilogram of body weight (gc/kg).
  Interventions: Genetic: CSL222 (Adeno-associated viral vector serotype 5 [AAV5]-hFIXco-Padua)

INTERVENTIONS:
Genetic: CSL222 (Adeno-associated viral vector serotype 5 [AAV5]-hFIXco-Padua) — Administered as a single IV infusion.
  Other Names: Etranacogene Dezaparvovec

SUMMARY:
This is a phase 3, prospective, open-label, single-arm, single-dose, multicenter study investigating the efficacy, safety, and tolerability of CSL222 (AAV5-hFIXco-Padua) in adolescent male participants with severe or moderately severe hemophilia B.

ELIGIBILITY:
Inclusion Criteria:

* Key Inclusion Criteria for the Lead-in Period:

Assigned male sex at birth

* Aged >=138 months (11 years and 6 months) to less than (<) 206 months (17 years and 2 months) at the time of informed consent / assent.
* Congenital hemophilia B with known severe or moderately severe FIX deficiency (less than or equal to [<=] 2% of normal circulating FIX) for which the participant has been on continuous FIX prophylaxis.
* On stable continuous FIX prophylaxis for at least 2 months before Screening.
* Minimum of 75 previous exposure days of treatment with FIX protein before Screening.
* Additional Key Inclusion Criteria for the Treatment Period:

Completed the Lead-in Period: minimum of 6 months (26 weeks) of lead-in data collected and eligibility has been confirmed.

* Aged >= 12 to < 18 years at the time of CSL222 treatment.

Exclusion Criteria:

* Key Exclusion Criteria for the Lead-in Period:

History of FIX inhibitors or positive FIX inhibitor test at Screening (based on central laboratory results).

* Screening laboratory values (based on central laboratory results):

  * Total bilirubin > 2 × the upper limit of normal (ULN).
  * Alanine aminotransferase (ALT) > 2 × the ULN.
  * Aspartate aminotransferase (AST) > 2 × the ULN.
  * Alkaline phosphatase (ALP) > 2 × the ULN.
  * Serum creatinine > 2 × the ULN.
  * Hemoglobin < 8 g/dL.
* Any condition other than hemophilia B resulting in an increased bleeding tendency.
* Thrombocytopenia, defined as a platelet count below 50 × 10^9/L, at screening (based on central laboratory results).
* Any uncontrolled or untreated infection (human immunodeficiency virus, hepatitis C, etc) or any other significant concurrent, uncontrolled medical condition, as evaluated by the investigator, including, but not limited to renal, hepatic, cardiovascular, hematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral, or psychiatric disease, alcoholism, drug dependency, or any other psychological disorder evaluated by the investigator to interfere with adherence to the Clinical Study Protocol procedures or with the degree of tolerance to CSL222.
* Additional Key Exclusion Criteria for the Treatment Period:

Positive FIX inhibitor test at Visit L-Final (based on central laboratory results)

* AAV5 NAb titer > 1:900 as assessed at Visit LX (last visit before Visit L-Final).
* Visit L-Final laboratory values (based on central laboratory results) of:

  * Total bilirubin > 2 × the ULN
  * ALT > 2 × the ULN.
  * AST > 2 × the ULN.
  * ALP > 2 × the ULN.
  * Serum creatinine > 2 × the ULN.
  * Hemoglobin < 8 g/dL.
* Thrombocytopenia, defined as a platelet count below 50 × 10^9/L, at Visit L-Final (based on central laboratory results).

Ages: 138 Months to 206 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Assigned male at birth.
Enrollment: 20 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2033-10-24 (Estimated); Study Completion 2033-10-24 (Estimated)

PRIMARY OUTCOMES:
Annualized Bleeding Rate (ABR) | For the Lead-In Period (at least 6 months) and for the 52 weeks after stable FIX expression (months 7 to 18 after treatment with CSL222)

SECONDARY OUTCOMES:
Canadian Hemophilia Outcomes-Kids Life Assessment Tool (CHO-KLAT) total score and change from baseline | At baseline and Month 18 post treatment
  The CHO-KLAT is designed to measure aspects of quality of life for boys with hemophilia. CHO-KLAT is a 40-item questionnaire, available in both child self-report (for ages 7 to 18) and parent-proxy versions (for ages 4 to 18). Items are categorized into 7 key domains (Activities, Autonomy, Bleeding, Emotional Health, Hemophilia Knowledge, Social Functioning, and Treatment). The measure is scored on a scale of 0 to 100, with 100 indicating best health-related quality of life.
Endogenous FIX activity | At baseline, and at months 6, 12, and 18 after treatment with CSL222
Change from baseline in endogenous FIX activity | At baseline, and at months 6, 12, and 18 after treatment with CSL222
Annualized consumption of FIX replacement therapy | For the Lead-In Period (at least 6 months), for the 52 weeks following stable FIX expression (months 7 to 18 after treatment with CSL222), and annually in the Posttreatment Follow-up Period (up to 5 years)
  Mean annualized consumption (IU/year) of FIX replacement therapy (excluding FIX replacement for invasive procedures).
Annualized infusion rate of FIX replacement therapy | For the Lead-In Period (at least 6 months), for the 52 weeks following stable FIX expression (months 7 to 18 after treatment with CSL222), and annually in the Posttreatment Follow-up Period (up to 5 years)
  Mean annualized infusion rate (infusions/year) of FIX replacement therapy (excluding FIX replacement for invasive procedures).
Number of participants remaining free of continuous FIX prophylaxis | During the 52 weeks after stable FIX expression (months 7 to 18 after treatment with CSL222), and during months 7 to: 24, 36, 48, and 60 after treatment with CSL222
Percentage of participants remaining free of continuous FIX prophylaxis | During the 52 weeks after stable FIX expression (months 7 to 18 after treatment with CSL222), and during months 7 to: 24, 36, 48, and 60 after treatment with CSL222
ABR for spontaneous, joint, and FIX-treated bleeding episodes | For the Lead-In Period (at least 6 months) and during the 52 weeks after stable FIX expression (months 7 to 18 after treatment with CSL222)
Correlation of FIX activity levels and pre-CSL222 AAV5 NAb titer | At the end of the Lead-in Period and during 6 to 18 months after treatment with CSL222
Number of new target joints and resolution of preexisting target joints | During the 52 weeks after stable FIX expression (months 7 to 18 after treatment with CSL222), and then annually during the Posttreatment Follow-up Period (up to 5 years)
Number of participants with zero bleeds and zero FIX-treated bleeds | During the 52 weeks after stable FIX expression (months 7 to 18 after treatment with CSL222), and during months 7 to: 24, 36, 48, and 60 after treatment with CSL222
Percentage of participants with zero bleeds and zero FIX-treated bleeds | During the 52 weeks after stable FIX expression (months 7 to 18 after treatment with CSL222), and during months 7 to: 24, 36, 48, and 60 after treatment with CSL222
Change in the EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) Visual Analogue Scale (VAS) Overall Score | At baseline, during the Lead-In Period (at least 6 months), and in the Posttreatment Follow-up Period (up to 5 years)
  The EQ-5D-5L questionnaire visual analogue scale (VAS) measures overall health status on a vertical VAS ranging from 0 to 100. A higher score indicates better quality of life. The change from baseline in the EQ-5D-5L VAS score will be determined.
Change in the EQ-5D-5L Index Scores | At baseline, during the Lead-In Period (at least 6 months), and in the Posttreatment Follow-up Period (up to 5 years)
  The EQ-5D-5L questionnaire descriptive system of health-related quality of life consists of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) for which responses will be recorded on 5 levels of severity (no problems, slight problems, moderate problems, severe problems, and extreme problems). The responses will be converted into a single index utility score (typically between -0.6 and 1). A higher score indicates better quality of life. The change from baseline in the EQ-5D-5L index score will be determined.
Change in the Patient-Reported Outcomes Measurement Information System (PROMIS)-25 total score | At baseline, during the Lead-In Period (at least 6 months), and in the Posttreatment Follow-up Period (up to 5 years)
  For participants of age 12-16 years. PROMIS-25 is a collection of short forms measuring quality of life in children. It includes domains of physical function mobility, anxiety, depression, fatigue, peer relationships, and pain interference. Each domain consists of 4 questions and are scored from 1 to 5. PROMIS-25 also includes one question on pain intensity that is available as a numeric rating scale and is scored from 0 (no pain) to 10 (worst imaginable pain).
Change from baseline in PROMIS-29 total score | At baseline, during the Lead-In Period (at least 6 months), and in the Posttreatment Follow-up Period (up to 5 years)
  For participants of age >=17 years. PROMIS-29 is a collection of short forms consisting of 7 PROMIS domains in depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability to participate in social roles and activities. Each domain consists of 4 questions and are scored from 1 to 5. PROMIS-29 also includes 1 question on pain intensity that is available as a numeric rating scale and is scored from 0 (no pain) to 10 (worst imaginable pain).
Number of participants with endogenous FIX activity of => 5% | Up to 5 years after treatment with CSL222
Percentage of participants with endogenous FIX activity of => 5% | Up to 5 years after treatment with CSL222
Adverse events - number of participants | During the Lead-in Period (at least 6 months) and during the Posttreatment Follow-up Period (up to 5 years).
Adverse events - percentage of participants | During the Lead-in Period (at least 6 months) and during the Posttreatment Follow-up Period (up to 5 years).
Adverse events - number of events | During the Lead-in Period (at least 6 months) and during the Posttreatment Follow-up Period (up to 5 years).
Change in liver ultrasound | At baseline, month 12 and every 6 months thereafter up to 5 years after CSL222 treatment
Number of participants with antibodies against AAV5 | From treatment with CSL222 through end of study (up to 5 years after treatment with CSL222)
Number of participants who develop FIX inhibitors | From treatment with CSL222 through end of study (up to 5 years after treatment with CSL222)
Number of clinically significant clinical laboratory tests (Hematology and Biochemistry) reported as an AE | At baseline and up to 5 years after treatment with CSL222
Number of participants with clinically significant ALT/AST levels | At baseline and up to 5 years after treatment with CSL222
Percentage of participants with clinically significant ALT/AST levels | At baseline and up to 5 years after treatment with CSL222
Number of participants using corticosteroid for change in AST/ALT levels | Up to 5 years after treatment with CSL222
Duration of corticosteroid use for change in AST/ALT levels | Up to 5 years after treatment with CSL222
Mean inflammatory markers values | Up to 5 years after treatment with CSL222
  Inflammatory markers include interleukin (IL) -1-beta, IL-2, IL-6, interferon-gamma, and monocyte chemoattractant protein-1 (MCP-1) will be measured and reported as picograms per milliliter (pg/mL).
Change from baseline in Inflammatory markers | At baseline and up to 5 years after treatment with CSL222
  Inflammatory markers include IL -1-beta, IL-2, IL-6, interferon-gamma, and MCP-1

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (7):
- United States (4):
  - University of Florida, Gainesville, Florida
  - Arthur M. Blank Hospital - Children's Healthcare of Atlanta, Atlanta, Georgia
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - St. Jude Children's Research Hospital, Memphis, Tennessee
- Chaim Sheba Medical Center, Ramat Gan, Israel
- United Kingdom (2):
  - St Thomas Hospital, London
  - John Radcliffe Hospital - Oxford University Hospitals NHS, Oxford

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (ie FDA, EMA) is complete and the primary publication is available.
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.